CLINICAL TRIAL: NCT03380182
Title: Acupuncture and Acupressure for Postoperative Nausea and Vomiting in Children Undergoing Outpatient Middle Ear Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 987983
Record Dates: First submitted 2017-11-28; First posted 2017-12-21 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Nausea; Vomiting; PONV
Keywords: acupuncture; acupressure
MeSH Terms: conditions — Nausea; Vomiting; Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture/Acupressure Group (Experimental): Bilateral P6 point acupuncture will be performed intra-operatively by the PI, who has UC Davis Medical Center privilege for this specific acupuncture, while the patient is under anesthesia. Patient will be sent home with an acupressure band, which is to remain on for 24 hours post operatively.
  Interventions: Other: Acupressure Band
- Control Group (Sham Comparator): Bilateral sham point acupuncture will be performed intra-operatively. Patient will be sent home with a wrist sham band matching in appearance of acupressure bands without the acupressure function, which is to remain on for 24 hours post operatively.
  Interventions: Other: Sham Band

INTERVENTIONS:
Other: Acupressure Band — These bands use pressure to stimulate the P6 acupuncture point.
  Arms: Acupuncture/Acupressure Group
Other: Sham Band — These sham bands are used to make it seem like the band is using pressure to stimulate the P6 acupuncture point.
  Arms: Control Group

SUMMARY:
The specific aim of this study is to determine the incidence of post-operative nausea and vomiting (PONV) in the pediatric population undergoing outpatient middle ear surgery.

DETAILED DESCRIPTION:
The specific aim of this study is to determine the incidence of post-operative nausea and vomiting (PONV) in the pediatric population undergoing outpatient middle ear surgery receiving our institution's standard dual prophylactic antiemetic therapy in combination with intraoperative acupuncture and postoperative acupressure compared to those receiving only the standard dual prophylactic antiemetic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy ASA 1 and 2 Patients
* Age 2 to 18 years old
* Undergoing Outpatient Middle ear surgery

Exclusion Criteria:

* ASA 3 and above
* Patients with underlying pro-emetogenic disease
* Patients currently taking antiemetic agents
* pregnant women
* Cognitively impaired adults
* prisoners
* History of bleeding disorder
* Age less than 2 or greater than 18

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
The evaluation of post operative nausea and vomiting at different time points during and after hospital stay. | 24 hours
  number of emesis events

SECONDARY OUTCOMES:
number of antiemetics administered during the study period, | 24 hrs
  number of antiemetics administered
time to oral intake tolerance | 24 hrs
  time measured in minutes
duration of recovery room stay | 24 hours
  time measured in minutes
nausea requiring admission to hospital, emergency room or another medical care providers | 24 hrs
  Desc: number of events requiring ER visit, hospitalization or care from another medical care provider

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No